CLINICAL TRIAL: NCT03528460
Title: Étude Des Facteurs prédictifs Des Effets Cliniques et Des Complications à Court et Long Terme de la Stimulation cérébrale Profonde Des Noyaux Sous-thalamiques Dans la Maladie de Parkinson
Brief Title: Predictive Factors of Short/Long-term Outcome and Complications of Bilateral DBS in PD
Acronym: PREDIMPSTIM
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.272; 2092048 (Other: CNIL)
Record Dates: First submitted 2017-11-14; First posted 2018-05-17 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Deep Brain Stimulation; Subthalamic Nucleus; Predictive factors
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose and main objective of this study is the research of pre-operative and operative predictive factors of short-term (1-year) and long-term (15-years) improvement of quality of life, motor and non-motor symptoms in Parkinson's disease patients who have undergone to bilateral Subthalamic Nucleus Deep Brain Stimulation.

The hypothesis of the study is that the definition of pre-operative and operative predictive factors could be able to improve the pre-operative prognostic accuracy of outcome and complications after surgery, allowing also a better selection of the most suitable candidates for bilateral Subthalamic Nucleus Deep Brain Stimulation.

For example, we can suppose that an older age at surgery, elevated axial score, a less preoperative dopa-responsiveness, the presence of mild executive dysfunction at surgery or an unfavourable social status, could negatively influence the short and long term surgery outcome

DETAILED DESCRIPTION:
Subthalamic NucleusDeep Brain Stimulation (STN-DBS) represents a short and long-term effective treatment in Parkinson's disease (PD) patients. Various randomized controlled trials have confirmed the superiority of STN-DBS compared to the best medical treatment in patients with advanced Parkinson disease in term of improvement of motor function and quality of life. On the other hand, STN- DBS is associated with an increased risk of adverse events compared to best medical treatment.

Data from previous meta-analysis have shown that only pre-operative dopa-responsiveness can predict the clinical efficacy and outcome of STN-DBS. In particular the improvement of STN-DBS on quality of life mainly concern the physical aspects of functioning with a lower improvement on social and cognitive aspects.

However, not all of PD symptoms respond similarly to STN-DBS. In particular the effects of STN-DBS on the so-called levodopa unresponsive symptoms (i.e. gait and balance symptoms, autonomic dysfunction, sleep disorders, cognitive decline and speech and swallowing troubles) are modest or absent. Furthermore, levodopa unresponsive symptoms are one of the main causes of impairment and disability in advanced PD patients. Bearing in mind these informations, the clinical phenotyping of candidates for surgery appear crucial for the prediction of DBS outcome and selection of better candidates. In the recent years, several papers highlighted and expanded the list of possible predictive factors, from a motor point of view to non-motor symptoms and psychosocial aspects.

In this setting, the aim of our study is to determine the pre-operative and operative short-term (1-year) and long-term (15-years) predictive factors of improvement of quality of life and motor and non-motor symptoms in a large cohort of PD patients who have undergone to bilateral STN-DBS. The better definition of short-term and long-term predictive factors and its association with the different PD different clinical phenotypes could allow in the future a better definition of the effects of STN-DBS on quality of life and motor and non-motor symptoms in the different PD clinical phenotypes.

In the same way, it could be assumed that a better definition of pre-operative predictive factors of surgical, hardware and stimulation-induced STN-DBS side effects in the short term, could also allow a better definition of the risk-to-benefit ratio and outcome after STN-DBS surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease treated with bilateral Subthalamic Nucleus Deep Brain Stimulation

Exclusion Criteria:

* Patients treated with bilateral Subthalamic Nucleus Deep Brain Stimulation not affected by Parkinson's Disease
* Patients with Parkinson's disease treated with unilateral Subthalamic Nucleus Deep Brain Stimulation

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Parkinson's disease treated with bilateral Subthalamic Nucleus Deep Brain Stimulation
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2019-01-27 (Actual)

PRIMARY OUTCOMES:
Changes in the Unified Parkinson's Disease Rating Scale (UPDRS) section I, II, III, IV, V, VI scores | pre-operative evaluation, 1-year and 15-years after Subthalamic Nucleus Deep Brain Stimulation
  The Unified Parkinson's Disease Rating Scale (UPDRS) has been developed for the clinical evaluation of Parkinson's disease (PD) patients. It allows the assessment of both motor and non-motor symptoms associated with PD

SECONDARY OUTCOMES:
Number of Patients that developed Treatment-Related (drug-related or DBS-related) complications | 1 year after bilateral Subthalamic Nucleus Deep Brain Stimulation
  Surgical-related complications, post-operative complications related to DBS devices and hardware, complications related to STN stimulation or drug administration.
  Post-operative complications directly related to STN stimulation.
Changes in the Parkinson's Disease Questionnaire (PDQ-39) total score and different subscale scores (Mobility; Activities of daily living; Emotional well being; Stigma; Social Support; Cognitions; Communication; Bodily discomfort) | pre-operative evaluation, 1-year and 15-years after Subthalamic Nucleus Deep Brain Stimulation
  The Parkinson's Disease Questionnaire (PDQ-39) is a short 39 item self-report health status questionnaire developed for evaluate the quality of life in Parkinson's disease patients.
Changes in the Movement Disorder Society (MDS)-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part I, II, III, IV scores | pre-operative evaluation, 1-year after Subthalamic Nucleus Deep Brain Stimulation
  The Movement Disorder Society (MDS)-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is the recent version of the UPDRS revised by the MDS. It allows the assessment of both motor and non-motor symptoms associated with PD

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cavallieri, MD, Principal Investigator — CHU Grenoble Alpes; Elena Moro, MD, PhD, Study Director — CHU Grenoble Alpes
Locations (1):
- Moro, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kleiner-Fisman G, Herzog J, Fisman DN, Tamma F, Lyons KE, Pahwa R, Lang AE, Deuschl G. Subthalamic nucleus deep brain stimulation: summary and meta-analysis of outcomes. Mov Disord. 2006 Jun;21 Suppl 14:S290-304. doi: 10.1002/mds.20962. PMID 16892449
- [Result] Weaver FM, Follett K, Stern M, Hur K, Harris C, Marks WJ Jr, Rothlind J, Sagher O, Reda D, Moy CS, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein J, Stoner G, Heemskerk J, Huang GD; CSP 468 Study Group. Bilateral deep brain stimulation vs best medical therapy for patients with advanced Parkinson disease: a randomized controlled trial. JAMA. 2009 Jan 7;301(1):63-73. doi: 10.1001/jama.2008.929. PMID 19126811
- [Result] Moro E, Lozano AM, Pollak P, Agid Y, Rehncrona S, Volkmann J, Kulisevsky J, Obeso JA, Albanese A, Hariz MI, Quinn NP, Speelman JD, Benabid AL, Fraix V, Mendes A, Welter ML, Houeto JL, Cornu P, Dormont D, Tornqvist AL, Ekberg R, Schnitzler A, Timmermann L, Wojtecki L, Gironell A, Rodriguez-Oroz MC, Guridi J, Bentivoglio AR, Contarino MF, Romito L, Scerrati M, Janssens M, Lang AE. Long-term results of a multicenter study on subthalamic and pallidal stimulation in Parkinson's disease. Mov Disord. 2010 Apr 15;25(5):578-86. doi: 10.1002/mds.22735. PMID 20213817
- [Result] Castrioto A, Lozano AM, Poon YY, Lang AE, Fallis M, Moro E. Ten-year outcome of subthalamic stimulation in Parkinson disease: a blinded evaluation. Arch Neurol. 2011 Dec;68(12):1550-6. doi: 10.1001/archneurol.2011.182. Epub 2011 Aug 8. PMID 21825213
- [Result] Guehl D, Cuny E, Benazzouz A, Rougier A, Tison F, Machado S, Grabot D, Gross C, Bioulac B, Burbaud P. Side-effects of subthalamic stimulation in Parkinson's disease: clinical evolution and predictive factors. Eur J Neurol. 2006 Sep;13(9):963-71. doi: 10.1111/j.1468-1331.2006.01405.x. PMID 16930362